CLINICAL TRIAL: NCT04789837
Title: The Phosphodiesterase 3 Inhibitor Cilostazol as an Adjunct to Conventional Therapy in Patients With Osteoarthritis: A Proof-of-Concept, Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: The Phosphodiesterase 3 Inhibitor Cilostazol as an Adjunct to Conventional Therapy in Patients With Osteoarthritis
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Institutional and funding constrains
Sponsor: Sadat City University (Other)
Responsible Party: Principal Investigator, Mahmoud Samy Abdallah, Principle Investigator, Sadat City University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15/2021RHU
Record Dates: First submitted 2021-03-06; First posted 2021-03-10 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Cilostazol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cilostazol (Experimental): Cilostazol 50 mg twice daily plus Celecoxib 200mg capsule
  Interventions: Drug: Cilostazol 50 MG
- Placebo (Placebo Comparator): Placebo tablet twice daily plus Celecoxib 200mg capsule
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cilostazol 50 MG — Cilostazol 50 mg twice daily plus Celecoxib 200mg capsule
  Arms: Cilostazol
Drug: Placebo — Placebo tablet twice daily plus Celecoxib 200mg capsule
  Arms: Placebo

SUMMARY:
Cilostazol is able to suppress the degradation of type II collagen in human chondrocytes induced by IL-1b. Cilostazol add-on for celecoxib therapy has synergistic anti-arthritic potential by inhibiting proinflammatory cytokine production in synovial fibroblasts through the IL-10/SOCS3 pathways, consequently leading to the inhibition of synovial cell proliferation and overcoming the perpetuation of synovial inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Primary osteoarthritis Patients recruited were between 30 to 60 years of age, with X-ray confirmed Kellgren-Lawrence grade13 II or III severity primary tibiofemoral OA, according to the American College of Rheumatology criteria.

Exclusion Criteria:

* Those patients were excluded from the present study who:

  * were of age less than 30 years or more than 60 years
  * presented with active concomitant gastroduodenal disorders, hepatic and renal impairment within last 30 days prior to receiving the study drug
  * were diagnosed to have any inflammatory arthritis, gout or acute trauma of the knee, hip or spine; accompanying OA of the hip of sufficient severity to interfere with the functional assessment of the knee
  * had previous or ongoing treatment with oral SYSDOA (e.g., glucosamine sulphate, chondroitin sulphate, diacerein, piascledine), anti-depressants, tranquillisers, antacids or antibiotics; were having active cardiac lesion or hypertension, were pregnant females and those who were planning their pregnancy during the study
  * were having a known hypersensitivity to the used medications
  * have persistent diarrhoea or laxative use; severe gastrointestinal disorders, severe obesity, severe parenchymal organ disease, or anaemia (haemoglobin< 10.0 g/ dl or haematocrit < 30%).
  * Patients who received oral, intramuscular, intraarticular or soft tissue injections of corticosteroids within last eight weeks before receiving the first dose of the study medication, or had undergone joint lavage and arthroscopic procedures in the previous 6 months, were also excluded.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue scale assessment of pain | week 12
  the change of Visual Analogue Scale (VAS) pain score from baseline to posttreatment. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain."

SECONDARY OUTCOMES:
WOMAC change | week 12
  the change of WOMAC Osteoarthritis Index from baseline to posttreatment
the change of Short Form 36 Questionnaire (SF-36) score from baseline to posttreatment | week 12
  The SF-36 is a generic instrument to assess health-related quality of life. It consists of 36 questions and assesses 8 dimensions: physical functioning, role physical, pain index, general health, vitality, social functioning, role emotional, and mental health index. It also provides 2 summary measures of physical and mental components. The SF-36 score ranges from 0 to 100, with higher scores indicating better health status.
Adverse drug reaction | 12 weeks
  Clinical side effects
Interleukin 1 beta | 12 weeks
  Interleukin 1 beta serum level
Serum level Tumor necrosis factor- alpha (TNF-α) | 12 weeks
  Serum level Tumor necrosis factor- alpha (TNF-α)
Serum levels of IL-17 | 12 weeks
  Serum levels of IL-17
Serum levels of BDNF | 12 weeks
  Serum levels of BDNF
Serum levels of IL-10 | 12 WEEKS
  Serum levels of IL-10

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Pharmacy, Shibīn al Kawm, Menoufia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF